CLINICAL TRIAL: NCT06781112
Title: Prospective, Single Center, Single Arm Phase II Clinical Study of TPF Combined With Immune Checkpoint Inhibitor Induction Therapy for Locally Advanced Nasopharyngeal Carcinoma Patients
Brief Title: A Phase II Study of TPF With PD-1 Inhibitor Induction Therapy for Locally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weiwei Zhang (Other)
Responsible Party: Sponsor-Investigator, Weiwei Zhang, Clinical Professor, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ethical2024-079(Science)-01; 2024276 (Other Grant/Funding Number: Chengdu Municipal Health Commission)
Record Dates: First submitted 2025-01-11; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: TPF; Immunotherapy; Nasopharyngeal Carcinoma; Phase II Clinical Study
Keywords: TPF; Immunotherapy; Nasopharyngeal Carcinoma; phase II clinical study
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil; tislelizumab; Therapeutics

STUDY DESIGN:
Intervention Model Description: TPF induction chemotherapy combined with tislelizumab+cisplatin concurrent chemoradiotherapy combined with tislelizumab adjuvant therapy (experimental group): TPF induction chemotherapy (albumin paclitaxel 200mg/m2+cisplatin 60mg/m2, divided into 3 days of infusion+5-fluorouracil 3000mg/m2, continuously intravenously pumped for 120 hours)+trastuzumab 200mg d1, once every 3 weeks, for a total of 3 courses+concurrent chemoradiotherapy combined with tislelizumab (cisplatin 100mg/m2+tislelizumab 200mg, starting from the first day of radiotherapy, once every 3 weeks during radiotherapy, for a total of 3 courses), synchronous IMRT+tislelizumab adjuvant therapy (tislelizumabb 200mg d1, once every 3 weeks) (8 trips in total)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPF combined with immunotherapy for LA-NPC (Experimental): Induction chemotherapy with PD-1 inhibitor combined with TPF (albumin paclitaxel, cisplatin and 5-fluorouracil) regimen, administered every 3 weeks: albumin paclitaxel (200mg/m2), cisplatin (60mg/m2, infused over 3 days), 5-fluorouracil (3000mg/m2, continuously intravenously pumped for 120 hours), and PD-1 inhibitor ( 200mg).All patients received 3 cycles of induction therapy followed by radical concurrent chemoradiotherapy combined with tislelizumab (200mg) treatment, Q3W. The cisplatin in the synchronous chemoradiotherapy regimen is administered once a week, with a dose of 40mg/m2 per dose, and the total dose of cisplatin does not exceed 100mg/m2. For patients who cannot tolerate cisplatin during synchronous radiotherapy and chemotherapy, cisplatin may not be combined.
  Interventions: Drug: albumin paclitaxel (200mg/m2), cisplatin (60mg/m2, infused over 3 days), 5-fluorouracil (3000mg/m2, continuously intravenously pumped for 120 hours), and tislelizumab ( 200mg).

INTERVENTIONS:
Drug: albumin paclitaxel (200mg/m2), cisplatin (60mg/m2, infused over 3 days), 5-fluorouracil (3000mg/m2, continuously intravenously pumped for 120 hours), and tislelizumab ( 200mg). — Induction chemotherapy with PD-1 inhibitor combined with TPF regimen, administered every 3 weeks: albumin paclitaxel (200mg/m2), cisplatin (60mg/m2, infused over 3 days), 5-fluorouracil (3000mg/m2, continuously intravenously pumped for 120 hours), and PD-1 inhibitor ( 200mg).
  All patients received 3 cycles of induction therapy followed by radical concurrent chemoradiotherapy combined with tislelizumab (200mg) treatment, Q3W. The cisplatin in the synchronous chemoradiotherapy regimen is administered once a week, with a dose of 40mg/m2 per dose, and the total dose of cisplatin does not exceed 100mg/m2. For patients who cannot tolerate cisplatin during synchronous radiotherapy and chemotherapy, cisplatin may not be combined.
  Other Names: radical concurrent chemoradiotherapy combined with tislelizumab (200mg) treatment

SUMMARY:
NPC is one of the most common malignant tumors in the head and neck region of China. Currently, the main treatment regimen for LA-NPC is radical concurrent chemoradiotherapy combined with induction or adjuvant chemotherapy. However, after radical radiotherapy and chemotherapy treatment, 15% -30% of patients still experience recurrence or distant metastasis. At present, the treatment options for R/M-NPC are very limited, especially for patients with recurrent or metastatic nasopharyngeal carcinoma who have failed second-line treatment, there is no standard treatment plan. Therefore, it is urgent to study a new treatment mode to improve the therapeutic efficacy of LA-NPC, thereby reducing the recurrence and metastasis rates.

This study explores the safety and efficacy of TPF combined with immune checkpoint inhibitor induction therapy in LA-NPC patients through prospective research. The results of this study are expected to provide new ideas and methods for the treatment of LA-NPC and provide reference for clinical practice. The investigators believe that induction chemotherapy combined with immunotherapy has broad application prospects in the field of LA-NPC, and is expected to bring better treatment effects and quality of life to patients, bringing new hope to the medical community and patients.

According to the inclusion criteria, eligible patients will be included:

Induction chemotherapy with Tislelizumab combined with TPF regimen, administered every 3 weeks: albumin paclitaxel (200mg/m2), cisplatin (60mg/m2, infused over 3 days), 5-fluorouracil (3000mg/m2, continuously intravenously pumped for 120 hours), and PD-1 inhibitor (Tislelizumab 200mg).

All patients received 3 cycles of induction therapy followed by radical concurrent chemoradiotherapy combined with Tislelizumab (200mg) treatment, Q3W. The cisplatin in the synchronous chemoradiotherapy regimen is administered once a week, with a dose of 40mg/m2 per dose, and the total dose of cisplatin does not exceed 100mg/m2. For patients who cannot tolerate cisplatin during synchronous radiotherapy and chemotherapy, cisplatin may not be combined. The IMRT radiotherapy area includes the primary tumor volume (GTVp), the total tumor volume of the affected lymph nodes (GTVn), the high-risk clinical target volume (CTV1), and the low-risk clinical target volume (CTV2). PTVp, PTV1, and PTV2 are respectively expanded by 3mm on GTVp, CTV1, and CTV2. The prescription doses for PTVp, PTVn, PTV1, and PTV2 are 70-72 Gy, 66-70 Gy, 60-68 Gy, and 54-58 Gy, respectively, with a total of 30-33 divided exposures.

After the completion of synchronous radiotherapy and chemotherapy, adjuvant therapy with Tislelizumab (Tislelizumab 200mg d1, once every 3 weeks, for a total of 8 courses) is administered. For patients with high-risk recurrence factors (T4 or N2), combination chemotherapy with capecitabine 625mg/m2 po bid is performed for one year.

Treat until any of the following conditions occur:

Disease progression; No clinical benefit; Intolerable toxicity; Withdrawal of informed consent; Or maintain treatment for up to six months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 75 years old, gender not limited;
2. Pathological diagnosis of nasopharyngeal non keratinizing carcinoma (differentiated or undifferentiated, i.e. WHO classification II or III);
3. Stage III-IVa (8th AJCC/UICC stage), excluding T3N0-1M0 patients;
4. Newly diagnosed nasopharyngeal carcinoma patients who have not received any anti-tumor treatment in the past;
5. The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) in the United States ranges from 0 to 1;
6. Having sufficient organ and bone marrow function, defined as follows:

   1. Blood routine: Neutrophil count (NEUT #) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 80 × 109/L; Hemoglobin ≥ 8 g/dL;
   2. Liver function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN); Total bilirubin (TBIL) ≤ 1.5 × ULN;
   3. Albumin ≥ 2.8 g/dL;
   4. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate (CCR)>60 ml/min;
   5. Coagulation function: International Normalized Ratio (INR) ≤ 1.5; Partial thromboplastin time (APTT) ≤ 1.5 × ULN;
7. The subjects voluntarily joined this study, signed an informed consent form, and were able to comply with the visit and related procedures specified in the protocol.

Exclusion Criteria:

1. Medical history of other malignancies (except for cured skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, gastrointestinal intramucosal carcinoma and other malignancies that the researchers think can be included);
2. Any active autoimmune disease or autoimmune disease history, including but not limited to immune related neurological disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue disease, scleroderma, inflammatory bowel disease, including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis (TEN) or Stevens Johnson syndrome (except for type I diabetes mellitus using a stable dose of insulin);
3. Individuals with allergic diseases, a history of severe drug allergies, and known allergies to any component of macromolecular protein preparations or PD-1 monoclonal antibody injections (note: severe allergies may result in hospitalization);
4. Received any of the following treatments:

   1. Patients who have previously used PD-1 antibody, PD-L1 antibody, PD-L2 antibody, CTLA-4 antibody;
   2. Individuals who have received anti-tumor vaccines;
   3. Use any active vaccine against infectious diseases (such as influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before the first administration or during the planned study period;
   4. Having undergone major surgery or suffered serious trauma within 4 weeks prior to the first administration of medication;
   5. The toxicity of previous anti-tumor treatments has not recovered to ≤ CTCAE 5.0 Grade 1 (excluding hair loss and sequelae related to previous platinum therapy neurotoxicity) or the level specified in the inclusion/exclusion criteria;
5. Patients with serious medical diseases, such as Grade II and above cardiac dysfunction (NYHA standard), ischemic heart disease (such as myocardial infarction or angina pectoris), clinically significant supraventricular or ventricular arrhythmia, poorly controlled diabetes (fasting blood glucose ≥ 10 mmol/L), poorly controlled hypertension (systolic blood pressure>150 mmHg and/or diastolic blood pressure>100 mmHg), and echocardiography showed ejection fraction<50%; QTc interval, male>450 milliseconds, female>470 milliseconds; Abnormal electrocardiogram examination and researchers believe there are additional risks to the investigational drug;
6. Subjects with a known history of interstitial pneumonia, a history of non infectious pneumonia, or a high suspicion of interstitial pneumonia; Or subjects who may interfere with the detection or treatment of suspected drug-related pulmonary toxicity; Allow subjects who have previously had drug-induced or radiation non infectious pneumonia but are asymptomatic to be included in the study; Individuals with active pulmonary tuberculosis or a history of tuberculosis infection that has not been controlled through treatment;
7. Patients with hyperthyroidism and organic thyroid disease cannot be included in the study. Hypothyroidism treated with stable doses of thyroid replacement hormone can be included, while hypothyroidism that can be controlled by thyroid replacement hormone treatment can be included (whether it can be controlled will be confirmed by the researcher and/or endocrinologist);
8. Presence of active infection, or unexplained fever occurring during screening or 48 hours prior to initial administration, or use of systemic antibiotics within one week prior to signing informed consent;
9. Active hepatitis B (HBV DNA ≥ 2000 IU/ml or 104 copies/ml) or hepatitis C (hepatitis C antibody positive, and HCV RNA higher than the detection limit of the analytical method), or a known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS);
10. Having a clear history of neurological or mental disorders, such as epilepsy or dementia;
11. Have a clear history of drug abuse or alcohol abuse within the past 3 months;
12. Pregnant or lactating women; The subjects (and their partners) have planned to have children, engaged in unprotected sexual activity, or are unwilling to use appropriate contraceptive measures (such as condoms, contraceptive rings, or partner sterilization) during the screening period until 3 months after the end of their study;
13. Received any investigational drug within 4 weeks prior to the first use of the investigational drug, or enrolled in another clinical study at the same time, unless it is an observational (non interventional) clinical study or an interventional clinical study follow-up;
14. The researchers determined that there may be other factors affecting the subjects in this study, which may prevent them from completing the trial medication and follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | From enrollment to the end of 3 cycles (each cycle is 21 days) introduction therapy
  Proportion of patients with complete remission (CR) and partial remission (PR)

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu University of Traditional Chinese Medicine Second Clinical School/Affiliated Chengdu Fifth People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Health Security Information Platform Medical Research Registration and Filing Information System — https://www.medicalresearch.org.cn/clinicalResearch/researchMain